CLINICAL TRIAL: NCT04339413
Title: An Open-Label, Multicenter, Rollover Study to Evaluate the Safety and Tolerability of Long-Term Administration of Gantenerumab in Participants With Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of Long-term Administration of Gantenerumab in Participants With Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate development of Gantenerumab for treatment of prodromal/mild/early stage Alzheimer's disease following results of a pre-planned analysis of the safety and efficacy of Gant in Graduate I&II (WN29922/WN39658).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WN41874
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCarlet RoAD (Experimental): Participants enrolled from the open label extension (OLE) part of parent study WN25203, received gantenerumab, up to 1200 milligram (mg), subcutaneous (SC) injection, every 4 weeks (Q4W) for up to 129 weeks.
  Interventions: Drug: Gantenerumab
- Marguerite RoAD (Experimental): Participants enrolled from the OLE part of parent study WN28745, received gantenerumab, up to 1200 mg, SC injection, Q4W for up to 129 weeks.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab was administered as SC injection Q4W.

SUMMARY:
The main purpose of the study was to evaluate the safety and tolerability of long-term administration of gantenerumab in participants with AD. All participants who have completed the open-label extensions (OLEs) of studies WN25203 or WN28745 were enrolled in Part 1 of this study. Of these, participants who completed Week 104 visit in Part 1. Participants received open-label gantenerumab by subcutaneous (SC) injection every four weeks (Q4W) at the same dose as administered in the parent studies (part 1)/ Week 104 visit.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Participants who completed the open-label extensions (OLEs) of studies WN25203 or WN28745 will be eligible to participate in Part 1 of the study
* Part 2: All participants who have completed Week 104 visit in Part 1 will be eligible for Part 2 of the study
* For Part 1 and Part 2:
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 16 weeks after the last dose of study drug
* Agreement to not donate blood or blood products for transfusion for the duration of the study and for 1 year after final dose of study drug
* Availability of a person ('caregiver') who in the investigator's judgement, has frequent and sufficient contact with the participant

Exclusion Criteria:

* Prematurely discontinued from the OLEs of studies WN25203 or WN28745 or from study drug for any reason
* Any medical condition that may jeopardize the participant's safety if he or she continues to receive study treatment
* If the participant is unlikely to benefit from gantenerumab therapy, based on disease progression or other factors, or if study participation is otherwise not in the participant's best interest
* Any investigational treatment other than gantenerumab during or since completion of the OLEs of studies WN25203 or WN28745
* Pregnancy
* Evidence of disseminated leptomeningeal hemosiderosis (i.e., more than three focal leptomeningeal hemosiderosis)
* Evidence of intracerebral macrohemorrhage
* Part 2: Participants who have been discontinued from Part 1 of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- United States (11):
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Accelerated Enrollment Solutions, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Bioclinica The Villages, The Villages, Florida
  - Western Michigan University Homer Stryker M.D. School of Medicine Center for Clinical Research, Kalamazoo, Michigan
  - Richmond Behavioral Associates, Staten Island, New York
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Central States Research, Tulsa, Oklahoma
  - Neurology Clinic PC, Cordova, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
- Instituto Neurologia Bs As, Ciudad Autonoma Buenos Aires, Argentina
- Australia (2):
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
- Canada (5):
  - Centricity Research, Halifax, Nova Scotia
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Alpha Recherche Clinique, Québec
- Especialidades Medicas LYS, Santiago, Chile
- Rigshospitalet, Hukommelsesklinikken, København Ø, Denmark
- Italy (5):
  - Nuovo Ospedale Civile S. Agostino-Estense; Clinica Neurologica ? Dipartimento di Neuroscienze, Modena, Emilia-Romagna
  - Azienda Ospedaliera Spedali Civili; Scienze Neurologiche, Brescia, Lombardy
  - IRCCS ?Centro S. Giovanni di Dio? Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - Irccs Multimedica Santa Maria; Unita' Di Neurologia, Castellanza, Lombardy
  - Fondazione San Raffaele Del Monte Tabor; Dipartimento Di Neurologia, Milan, Lombardy
- Japan (3):
  - Medical Corporation Hakuyokai Kashiwado Hospital, Chiba
  - Juntendo University Urayasu Hospital; Neurology, Chiba
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
- Mexico (3):
  - Hospital Mexico Americano, Guadalajara, Mexico CITY (federal District)
  - Hospital Universitario; Dr. Jose E. Gonzalez, Monterrey, Nuevo León
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
- Brain Research Center B.V, Amsterdam, Netherlands
- Poland (3):
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Późna
  - Przychodnia Specjalistyczna PROSEN, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
- Russia (2):
  - Saint Petersburg State Institution of Healthcare City Geriatric Medico-Social Center, Saint Petersburg, Sankt-Peterburg
  - FSMEI HPE ?Military Medical Academy n.a. S.M.Kirov"of Minist, Saint Petersburg, Sankt-Peterburg
- South Korea (3):
  - Inha University Hospital, Incheon
  - Seoul St Mary's Hospital, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
- Spain (7):
  - Hospital General Universitario de Elche; Servicio de Neurología, Elche, Alicante
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Fundación ACE; Servicio de Neurología, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
- Felix Platter-Spital Medizin Geriatrie, Basel, Switzerland
- Turkey (Türkiye) (3):
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Dokuz Eylul University Medicine Faculty; Noroloji Departmani, Izmir
  - Ondokuz Mayis University School of Medicine; Neurology, Samsun
- United Kingdom (4):
  - Llandough Hospital; Llandough Hospital Memory Team 3rd Floor Academic Building, Cardiff
  - Imperial Memory Unit, Charing Cross Hospital; Level 10 West, Department of Neurosciences, London
  - Campus for Ageing & Vitality; Clincal Ageing Research Unit, Newcastle
  - Hollins Park Hospital, Warrington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in Part 1 of the study at 56 centers in the United States, Spain, Canada, Italy, Germany, Japan, Korea, Mexico, Poland, Turkey, Australia, Russia, Argentina, Switzerland, Chile, Denmark, and Netherlands from 22 May 2020 to 04 Jan 2023. The study was terminated before Part 2 was initiated.
Pre-assignment Details: A total of 116 participants rolled over in this study of which 115 participants received gantenerumab in part 1. 59 participants rolled over from OLE WN25203 & 56 participants rolled over from WN28745. Due to negative pre-planned analysis of studies WN39658 & WN29922, this study was terminated by sponsor, & no participant was rolled over to Part 2.
Period: Overall Study
Arm/Group | SCarlet RoAD | Marguerite RoAD
Started | 59 | 57
Safety Evaluable Population (Safety evaluable population included all the participants who received at least one dose of gantenerumab) | 59 | 56
Completed | 1 | 0
Not Completed | 58 | 57
Not completed — Reason Not Specified | 2 | 7
Not completed — Study Terminated by Sponsor | 30 | 33
Not completed — Progressive Disease | 9 | 6
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Physician Decision | 3 | 1
Not completed — Death | 2 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all the participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | SCarlet RoAD | Marguerite RoAD | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (6.7) | 75.2 (8.3) | 76.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 13 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 56 | 42 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with gantenerumab and which does not necessarily have a causal relationship with gantenerumab. A Serious Adverse Event (SAE) is any significant hazard, contraindication, side effect that is fatal or life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is medically significant or requires intervention to prevent one or other of the outcomes listed above, and which does not necessarily have a causal relationship with gantenerumab.
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants
  AE | 54 | 49
  SAE | 11 | 10

2. Primary Outcome: Number of Participants With Change in Any Suicidal Ideation or Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of a participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, & attempts with actual/potential lethality. Categories have binary responses (yes/no) & include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0= no suicide risk present. Score of 1 or higher= suicidal ideation/behavior. Number of participants with any suicidal ideation/behavior were reported.
Time Frame: Baseline (Day 1), up to Week 104
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 56 | 54
Participants
  Baseline | 3 | 0
  Week 24: number analyzed (Participants) | 52 | 44
  Week 24 | 2 | 0
  Week 52: number analyzed (Participants) | 48 | 38
  Week 52 | 1 | 0
  Week 76: number analyzed (Participants) | 37 | 32
  Week 76 | 0 | 1
  Week 104: number analyzed (Participants) | 30 | 0
  Week 104 | 0 | 0

3. Primary Outcome: Number of Participants With Amyloid-Related Imaging Abnormalities-Edema (ARIA-E) AEs
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Amyloid-Related Imaging Abnormalities-Haemosiderin Deposition (ARIA-H) AEs
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Anti-drug Antibody (ADA) to Gantenerumab
Time Frame: Up to Week 133
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants | 3 | 1

6. Primary Outcome: Number of Participants With Injection-Site Reactions
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants | 14 | 7

7. Primary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered with gantenerumab and which does not necessarily have a causal relationship with gantenerumab. SAE is any significant hazard, contraindication, side effect that is fatal or life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is medically significant or requires intervention to prevent one or other of the outcomes listed above, and which does not necessarily have a causal relationship with gantenerumab.
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Population: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Measure: Count of Participants; unit: Participants
Arm/Group | SCarlet RoAD | Marguerite RoAD
Number analyzed (Participants) | 59 | 56
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Baseline [Day 1] up to 4 weeks after the last dose of study drug (Up to Week 133)
Description: Safety evaluable population included all the participants who received at least one dose of gantenerumab.
Groups:
- SCarlet RoAD: Participants enrolled from the OLE part of parent study WN25203, received gantenerumab, up to 1200 mg, SC injection, Q4W for up to 129 weeks.
Arm/Group | SCarlet RoAD | Marguerite RoAD
All-Cause Mortality (participants affected / at risk) | 2/59 | 0/56
Serious Adverse Events (participants affected / at risk) | 11/59 | 10/56
Other Adverse Events (participants affected / at risk) | 43/59 | 39/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCarlet RoAD (N=59) | Marguerite RoAD (N=56)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Death (General disorders) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCarlet RoAD (N=59) | Marguerite RoAD (N=56)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 3 (5)
Injection site reaction (General disorders) | 14 (183) | 7 (34)
Pyrexia (General disorders) | 1 (1) | 3 (4)
COVID-19 (Infections and infestations) | 13 (14) | 10 (10)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (12) | 7 (10)
Fall (Injury, poisoning and procedural complications) | 13 (20) | 8 (15)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Agitation (Psychiatric disorders) | 5 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04339413/Prot_SAP_000.pdf